CLINICAL TRIAL: NCT00044655
Title: Effectiveness of Switching Antipsychotic Medications
Brief Title: Switching Medication to Treat Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 98-924; R01MH059312 (NIH)
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Olanzapine; ziprasidone; Quetiapine Fumarate; Aripiprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stay on baseline medication prescribed (Active Comparator): Participants will continue taking medication prescribed at study entry: 1) either long-acting injectable haloperidol or fluphenazine, OR 2) two antipsychotic medications which might include a combination of any of the following: risperidone, olanzapine, ziprasidone, quetiapine, aripiprazole, or conventional (typical) antipsychotic medications.
  Interventions: Drug: Risperidone; Drug: Olanzapine; Drug: Ziprasidone; Drug: Quetiapine; Drug: Aripiprazole
- Switch per study protocol (Active Comparator): Participants will change medications from medication prescribed at study entry, either: 1) long-acting injectable risperidone, OR 2) one of the two antipsychotic medications prescribed at baseline which may include any of the following: risperidone, olanzapine, ziprasidone, quetiapine, aripiprazole, or conventional (typical) antipsychotic medications.
  Interventions: Drug: Risperidone; Drug: Olanzapine; Drug: Ziprasidone; Drug: Quetiapine; Drug: Aripiprazole

INTERVENTIONS:
Drug: Risperidone — As prescribed by routine prescriber (not dictated by study protocol)
  Other Names: Risperdal, Risperdal Consta
Drug: Olanzapine — As prescribed by routine prescriber (not dictated by study protocol)
  Other Names: Zyprexa
Drug: Ziprasidone — As prescribed by routine prescriber (not dictated by study protocol)
  Other Names: Geodon
Drug: Quetiapine — As prescribed by routine prescriber (not dictated by study protocol)
  Other Names: Seroquel
Drug: Aripiprazole — As prescribed by routine prescriber (not dictated by study protocol)
  Other Names: Abilify

SUMMARY:
This study will evaluate the effectiveness of switching medications in decreasing schizophrenia symptoms in individuals who are currently taking an antipsychotic medication for the treatment of schizophrenia.

DETAILED DESCRIPTION:
Over the past several years, new, "atypical" antipsychotic medications have become available to treat schizophrenia with little information to guide prescribing for relatively stable outpatients.

Participants will be randomly assigned to either continue taking their current medications for schizophrenia, or to switch to a new medication. Participants assigned to switch to a new medication will begin receiving either olanzapine (Zyprexa), risperidone (Risperdal), ziprasidone (Geodon), quetiapine (Seroquel), or aripiprazole (Abilify), depending on what they are currently taking. Participants currently taking a single oral medication will switch to olanzapine, risperidone, ziprasidone, quetiapine, or aripiprazole. Participants currently taking a single conventional injectable will begin taking long-acting injectable risperidone (Risperdal Consta). Participants currently taking two antipsychotic medications will begin taking only one of the medications they are currently using. Participants will stay on their assigned treatment for 6 months, after which time the participant's prescribing psychiatrist will advise the participant on which medication should be used. Study participants are interviewed at study start and at follow-up visits for 1 year.

ELIGIBILITY:
Inclusion criteria:

* SCID diagnosis of schizophrenia or schizoaffective disorder
* Partially remitted outpatients, defined as persons who have received clear symptomatic benefit from antipsychotic medication but remain symptomatic (due to lack of efficacy or inability to tolerate an efficacious dose) or suffer significant side effects
* Treatment with antipsychotic medications for at least 2 months
* Received at least 1 outpatient mental health service every 3 months for the past 6 months

Exclusion criteria:

* Severe symptoms or side effects that indicate the necessity for a medication change
* Currently taking 3 or more antipsychotic medications for ongoing daily administration (PRN medications and mood stabilizers are allowable)
* Treatment with clozapine
* One or more nights spent in a psychiatric hospitalization within the past 3 months
* Received services from a crisis intervention program within the past 3 months
* Require placement in a skilled nursing facility as a result of a physical condition or disability
* Criminal charges pending (once charges clear, the person will be considered)
* Pregnant or breast feeding
* Contraindication to any of the medications to which the patient might be assigned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2001-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Essock, PhD, Study Chair — Columbia University

REFERENCES:
- [Result] Covell NH, McEvoy JP, Schooler NR, Stroup TS, Jackson CT, Rojas IA, Essock SM; Schizophrenia Trials Network. Effectiveness of switching from long-acting injectable fluphenazine or haloperidol decanoate to long-acting injectable risperidone microspheres: an open-label, randomized controlled trial. J Clin Psychiatry. 2012 May;73(5):669-75. doi: 10.4088/JCP.11m07074. Epub 2012 Mar 6. PMID 22480442
- [Result] Essock SM, Schooler NR, Stroup TS, McEvoy JP, Rojas I, Jackson C, Covell NH; Schizophrenia Trials Network. Effectiveness of switching from antipsychotic polypharmacy to monotherapy. Am J Psychiatry. 2011 Jul;168(7):702-8. doi: 10.1176/appi.ajp.2011.10060908. Epub 2011 May 2. PMID 21536693

RESULTS

PARTICIPANT FLOW:
Groups:
- Stay: Participants will continue taking medication prescribed at study entry
- Switch: Participants will change medications from medication prescribed at study entry
Period: Overall Study
Arm/Group | Stay | Switch
Started | 102 | 117
Completed | 82 | 79
Not Completed | 20 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stay | Switch | Total
Number analyzed (Participants) | 102 | 117 | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 112 | 208
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (10.4) | 47.7 (11.3) | 46.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 31 | 73
  Male | 60 | 86 | 146
Region of Enrollment [Number; unit: participants]
  United States | 102 | 117 | 219

OUTCOME MEASURES:

1. Primary Outcome: Number Who Discontinued Medication Within First 6 Study Months
Time Frame: Measured at Six Months
Population: intent to treat samples for 2 substudies: injectable to injectable and polypharmacy to monotherapy
Measure: Number; unit: participants
Arm/Group | Stay | Switch
Number analyzed (Participants) | 92 | 97
participants | 11 | 23

2. Secondary Outcome: Psychiatric Symptoms, Hospitalization, and Medication Side Effects
Time Frame: Measured at Year 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Stay | Switch
Serious Adverse Events (participants affected / at risk) | 0/102 | 2/117
Other Adverse Events (participants affected / at risk) | 0/102 | 0/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stay (N=102) | Switch (N=117)
Psychiatric Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Following medication change, participant's prescriber called Project Director to report that the participant was not doing well and was hospitalized subsequent to symptom exacerbation; prescriber changed client's antipsychotic medication regime.
Death (Cardiac disorders) | 0 (0) | 1 (1) — Site PI learned that the 69 year old participant had died following recurrent episodes of bleeding from cerebral aneurism that was diagnosed, but unknown to the site PI, prior to study enrollment (randomized to injectable risperidone)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No